CLINICAL TRIAL: NCT01466673
Title: Comparative Study of the Effect on Acne With Norgestimate Containing Triphasic Oral Contraceptive and Biphasic Preparation Containing Desogestrel
Brief Title: An Efficacy and Safety Study Comparing Oral Contraceptive Containing Norgestimate or Desogestrel for Acne Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR015448; NRGMONCON4003
Record Dates: First submitted 2011-10-24; First posted 2011-11-08 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Ethinyl estradiol; Norgestimate; Desogestrel; Tricilest; Oilezz
MeSH Terms: conditions — Acne Vulgaris | interventions — Ethinyl Estradiol; norgestimate; Desogestrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ethinyl estradiol/Norgestimate (EE/NGM) (Experimental)
  Interventions: Drug: Ethinyl estradiol/Norgestimate (EE/NGM)
- Ethinyl estradiol/Desogestrel (EE/DSG) (Active Comparator)
  Interventions: Drug: Ethinyl estradiol/Desogestrel (EE/DSG)

INTERVENTIONS:
Drug: Ethinyl estradiol/Norgestimate (EE/NGM) — Ethinyl estradiol/Norgestimate encapsulated oral tablet will be administered once daily at bed time as 0.035/0.18 milligram (mg) for Days 1-7, 0.035/0.215 mg for Days 8-14, and 0.035/0.250 mg for Days 15-21 of EE/NGM, respectively up to 6 consecutive menstrual cycles consisting of 21 days each.
  Other Names: Tricilest
  Arms: Ethinyl estradiol/Norgestimate (EE/NGM)
Drug: Ethinyl estradiol/Desogestrel (EE/DSG) — Ethinyl estradiol/Desogestrel oral formulation will be administered once daily at bed time as 0.040/0.025 mg for Days 1-7, 0.030/0.125 mg for Days 8-22 of EE/DSG, respectively up to 6 consecutive menstrual cycles consisting of 22 days each.
  Other Names: Oilezz
  Arms: Ethinyl estradiol/Desogestrel (EE/DSG)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ethinyl estradiol and Norgestimate (EE/NGM) compared to Ethinyl estradiol and Desogestrel (EE/DSG), for treatment of female participants with mild to moderate acne vulgaris (pimples).

DETAILED DESCRIPTION:
This is a single-blind (physician does not know the name of the assigned drug) and randomized (study drug assigned by chance) study to compare the effectiveness and safety of EE/NGM and EE/DSG in female participants using oral contraceptive and have mild to moderate acne vulgaris. Tablets of EE/NGM and EE/DSG will be administered orally once daily for 6 months and will be instructed to visit for evaluation at Month 1, 3 and 6 post-administration. The efficacy will be evaluated efficacy primarily through total acne lesions count, which will be recorded at these evaluation visits. Unused study medications will be collected and drug accountability will be documented. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Needs contraception in the family planning - Mild to moderate acne vulgaris - Agrees to take only the supplied study drug as treatment for acne during the 6-month treatment phase of the study - Signs and dates an informed consent to participate in the study - female participants aged 18 to 45 years Exclusion Criteria: - Pregnant or nursing - Known hypersensitivity to any of the ingredients and currently having significant adverse experiences from ethinyl estradiol, norgestimate or desogestrel - Any coexisting medical condition or were taking any concomitant medication that is likely to interfere with safe administration of ethinyl estradiol/norgestimate and ethinyl estradiol/desogestrel, in the Investigator's opinion - Taking system retinoids, systemic antimicrobials, and topical acne treatments within 6 months, 1 month, and 2 weeks prior to enrollment, respectively - Taking investigational medication or oral contraceptives within 30 days prior to Screening

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd., Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (3):
- Thailand (3):
  - Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University, Bangkok
  - Department of Obstetrics and Gynecology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Department of Obstetrics and Gynecology, Faculty of Medicine, Chiang Mai University, Chiang Mai

REFERENCES:
- [Derived] Jaisamrarn U, Chaovisitsaree S, Angsuwathana S, Nerapusee O. A comparison of multiphasic oral contraceptives containing norgestimate or desogestrel in acne treatment: a randomized trial. Contraception. 2014 Nov;90(5):535-41. doi: 10.1016/j.contraception.2014.06.002. Epub 2014 Jun 12. PMID 25074072

RESULTS

PARTICIPANT FLOW:
Groups:
- Ethinyl Estradiol/Norgestimate (EE/NGM): Ethinyl estradiol/Norgestimate encapsulated oral tablet was administered once daily at bed time as 0.035/0.18 milligram (mg) for Days 1-7, 0.035/0.215 mg for Days 8-14, and 0.035/0.250 mg for Days 15-21 of EE/NGM, respectively up to 6 consecutive menstrual cycles consisting of 21 days each.
- Ethinyl Estradiol/Desogestrel (EE/DSG): Ethinyl estradiol/Desogestrel oral formulation was administered once daily at bed time as 0.040/0.025 mg for Days 1-7, 0.030/0.125 mg for Days 8-22 of EE/DSG, respectively up to 6 consecutive menstrual cycles consisting of 22 days each.
Period: Overall Study
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Started | 100 | 101
Completed | 93 | 95
Not Completed | 7 | 6
Not completed — Non-compliance with study treatment | 2 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG) | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Customized [Number; unit: Participants]
  Less than and equal to 18 years | 0 | 0 | 0
  Between 18 and 45 years | 100 | 101 | 201
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 101 | 201
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total and Each Type of Acne Lesions Count at Month 1
Description: Total acne (pimples) lesion (abnormal area of tissue, such as a wound, sore, rash, or boil) count is summation of all lesions which includes all comedones (open and closed), papules, pustules, and nodules. Change from Baseline means lesions at Baseline minus lesions at Month 1. Positive value indicates decrease in lesion count while negative value indicates increase in lesion count.
Time Frame: Baseline and Month 1
Population: Intent-to-treat population (ITT) included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Lesions
  Comedones Counts: Baseline | 10.97 (6.45) | 11.43 (7.58)
  Papules Counts: Baseline | 4.32 (4.94) | 4.46 (5.06)
  Pustules Counts: Baseline | 0.90 (1.96) | 1.12 (2.26)
  Nodules Counts: Baseline | 0.12 (0.86) | 0.00 (0.00)
  Total Counts: Baseline | 16.31 (9.57) | 17.00 (10.41)
  Comedones Counts: Change at Month 1 | 3.43 (4.82) | 3.44 (5.31)
  Papules Counts: Change at Month 1 | 0.20 (3.73) | 0.62 (2.19)
  Pustules Counts: Change at Month 1 | 0.35 (0.96) | 0.18 (0.82)
  Nodules Counts: Change at Month 1 | 0.12 (0.86) | -0.02 (0.20)
  Total Counts: Change at Month 1 | 4.10 (4.89) | 4.22 (5.91)

2. Primary Outcome: Change From Baseline in Total and Each Type of Acne Lesions Count at Month 3
Description: Total acne (pimples) lesion (abnormal area of tissue, such as a wound, sore, rash, or boil) count is summation of all lesions which includes all comedones (open and closed), papules, pustules, and nodules. Change from Baseline means lesions at Baseline minus lesions at Month 3. Positive value indicates decrease in lesion count while negative value indicates increase in lesion count.
Time Frame: Baseline and Month 3
Population: ITT population included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Lesions
  Comedones Counts: Change at Month 3 (n=93, 96) | 5.71 (6.93) | 5.60 (6.70)
  Papules Counts: Change at Month 3 (n=93, 96) | 2.83 (3.80) | 1.89 (2.92)
  Pustules Counts: Change at Month 3 (n=93, 96) | 0.63 (1.58) | 0.70 (1.50)
  Nodules Counts: Change at Month 3 (n=93, 96) | 0.12 (0.90) | 0.00 (0.00)
  Total Counts: Change at Month 3 (n=93, 96) | 8.84 (8.13) | 8.19 (7.78)

3. Primary Outcome: Change From Baseline in Total and Each Type of Acne Lesions Count at Month 6
Description: Total acne (pimples) lesion (abnormal area of tissue, such as a wound, sore, rash, or boil) count is summation of all lesions which includes all comedones (open and closed), papules, pustules, and nodules. Change from Baseline means lesions at Baseline minus lesions at Month 6. Positive value indicates decrease in lesion count while negative value indicates increase in lesion count.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Lesions
  Comedones Counts: Change at Month 6 (n=93, 95) | 9.02 (6.30) | 8.21 (7.43)
  Papules Counts: Change at Month 6 (n=93, 95) | 3.52 (5.08) | 2.77 (4.62)
  Pustules Counts: Change at Month 6 (n=93, 95) | 0.77 (2.17) | 0.96 (2.12)
  Nodules Counts: Change at Month 6 (n=93, 95) | 0.13 (0.89) | 0.00 (0.00)
  Total Counts: Change at Month 6 (n=93, 95) | 13.44 (9.74) | 11.94 (10.08)

4. Secondary Outcome: Number of Participants With Abnormal Vaginal Blood Loss at Month 1, 3 and 6
Description: Vaginal blood loss encompasses spotting and bleeding. Spotting is defined as a bleeding requiring no or at most one sanitary pad per day; however, bleeding requires two or more sanitary pads per day.
Time Frame: Month 1, 3 and 6
Population: Safety population included all randomized participants who received at least one dose of study medication. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Number; unit: Participants
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Participants
  Spotting at Month 1 (n=100,101) | 5 | 2
  Spotting at Month 3 (n=93, 96) | 6 | 4
  Spotting at Month 6 (n=93, 95) | 4 | 3
  Bleeding at Month 1 (n=100,101) | 13 | 4
  Bleeding at Month 3 (n=93, 96) | 4 | 7
  Bleeding at Month 6 (n=93, 95) | 6 | 3

5. Secondary Outcome: Number of Participants Non-Compliant With Therapy
Description: Compliance was assessed by transforming the data of forgotten tablets listed in the diary cards. Number of participants who forgot to take the drug was reported.
Time Frame: Month 1, 3 and 6
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Participants
  At Month 1 (n=100, 101) | 7 | 5
  At Month 3 (n=93, 96) | 13 | 10
  At Month 6 (n=93, 95) | 10 | 6

6. Secondary Outcome: Percentage of Participants With Categorical Score for Sebum Assessment at Month 1, 3 and 6
Description: Sebum assessment that is facial seborrhea (very oily skin) was assessed using sebutape strip on the forehead. Percentage of participants with facial seborrhea were assessed using categorical scores ranging from level 1 (lowest) to level 5 (highest). Highest level indicates worsening.
Time Frame: Baseline and Month 1, 3 and 6
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Percentage of Participants
  Level 1: Baseline (n=100,101) | 3.00 | 3.96
  Level 2: Baseline (n=100,101) | 10.00 | 12.87
  Level 3: Baseline (n=100,101) | 43.00 | 44.55
  Level 4: Baseline (n=100,101) | 31.00 | 34.65
  Level 5: Baseline (n=100,101) | 13.00 | 3.96
  Level 1: Month 1 (n=100,101) | 7.00 | 8.91
  Level 2: Month 1 (n=100,101) | 13.00 | 11.88
  Level 3: Month 1 (n=100,101) | 47.00 | 45.54
  Level 4: Month 1 (n=100,101) | 30.00 | 32.67
  Level 5: Month 1 (n=100,101) | 3.00 | 0.99
  Level 1: Month 3 (n=93, 96) | 6.45 | 10.42
  Level 2: Month 3 (n=93, 96) | 34.41 | 14.58
  Level 3: Month 3 (n=93, 96) | 45.16 | 59.38
  Level 4: Month 3 (n=93, 96) | 11.83 | 14.58
  Level 5: Month 3 (n=93, 96) | 2.15 | 1.04
  Level 1: Month 6 (n=93, 95) | 44.09 | 22.11
  Level 2: Month 6 (n=93, 95) | 27.96 | 43.16
  Level 3: Month 6 (n=93, 95) | 20.43 | 29.47
  Level 4: Month 6 (n=93, 95) | 6.45 | 5.26
  Level 5: Month 6 (n=93, 95) | 1.08 | 0.00

7. Secondary Outcome: Percentage of Participants Showing Treatment Response on the Investigator's Global Assessment at Month 6
Description: Percentage of participants showing treatment response on the Investigator's global assessment was graded on a 5-point scale as 0=worse, 1=no change, 2=fair, 3=good, and 4=excellent.
Time Frame: Month 6
Population: ITT population included all randomized participants who received at least one dose of study medication and fulfilled all inclusion and exclusion criteria. "N" signifies those participants who were evaluated for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 93 | 95
Percentage of participants
  0 (Worse) | 5.05 | 1.03
  1 (No Change) | 4.04 | 1.03
  2 (Fair) | 4.04 | 23.71
  3 (Good) | 43.43 | 52.58
  4 (Excellent) | 43.43 | 21.65

8. Secondary Outcome: Number of Participants With Treatment Response at the End-of-Therapy by Participant's Self-Assessment at Month 6
Description: Participant's self-assessment at end-of-therapy was measured by using the self-assessment questionnaire which included 3 questions, about the rating of acne improvement since start of study; comparison of this acne treatment with the one used in past and the continuity of treatment on physician's prescription to evaluate efficacy and acceptability of the study medication. The score was graded at 4 parameters as excellent, better, no change and worse.
Time Frame: Month 6
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 93 | 95
Participants
  Excellent | 47 | 35
  Better | 45 | 58
  No Change | 3 | 3
  Worse | 4 | 1

9. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Month 6
Description: Blood pressure is the pressure of blood flowing through blood vessels. Change from Baseline in blood pressure is the value at Month 6 minus value at Baseline.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Millimeters of Mercury
  Systolic BP: Baseline (n=100/101) | 110.6 (9.93) | 110.2 (10.61)
  Diastolic BP: Baseline (n=100/101) | 70.23 (8.08) | 69.47 (8.54)
  Systolic BP: Change at Month 6 (n=93, 95) | 0.33 (6.77) | -0.24 (8.98)
  Diastolic BP: Change at Month 6 (n=93, 95) | -0.80 (6.69) | -0.48 (7.76)

10. Secondary Outcome: Change From Baseline in Body Weight at Month 6
Description: Change from Baseline in body weight is the value at Month 6 minus value at Baseline.
Time Frame: Baseline and Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Number analyzed (Participants) | 100 | 101
Kilograms
  Baseline (n=100,101) | 55.62 (8.92) | 54.24 (9.36)
  Change at Month 6 (n=93,95) | -0.08 (1.89) | -0.20 (2.53)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Ethinyl Estradiol/Norgestimate (EE/NGM) | Ethinyl Estradiol/Desogestrel (EE/DSG)
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/101
Other Adverse Events (participants affected / at risk) | 34/100 | 60/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethinyl Estradiol/Norgestimate (EE/NGM) (N=100) | Ethinyl Estradiol/Desogestrel (EE/DSG) (N=101)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sudden severe headache (Nervous system disorders) | 1 (1) | 0 (0)
Dengue Hemorrhagic fever (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ethinyl Estradiol/Norgestimate (EE/NGM) (N=100) | Ethinyl Estradiol/Desogestrel (EE/DSG) (N=101)
Nausea (Gastrointestinal disorders) | 13 | 27
Vomiting (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 10
Somnolence (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 5 | 9
Libido increased (Reproductive system and breast disorders) | 0 | 2
Galactorrhoea (Reproductive system and breast disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Institution & Principal Investigator wish to publish information from Clinical Trial, a copy of manuscript must be provided to Sponsor at least 60 days prior to submission for publication/presentation and will arrange expedited reviews for the same. No paper with confidential information will be submitted without Sponsor's prior consent. If requested, Institution and Principal Investigator will hold such publication for up to additional 60 days to allow filing of patent application.